CLINICAL TRIAL: NCT00920842
Title: Metabolic Syndrome Following Transplant for Leukemia
Brief Title: Study of Metabolic Syndrome in Adolescent and Young Adult Survivors of Childhood Leukemia Who Have Undergone Stem Cell Transplant
Status: Completed | Type: Observational
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: K. S. Baker, MD, MS, Fred Hutchinson Cancer Research Center
Other Study IDs: IR 7141; P30CA077598 (NIH); UMN-2003NT063; CDR0000642276 (Registry Identifier: NCI); IR-6980 (Other: Former FHCRC IRB ID); FHCRC-2357.00 (Other: Former FHCRC ID)
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Cardiovascular Complications; Leukemia; Long-term Effects Secondary to Cancer Therapy in Children; Metabolic Syndrome
Keywords: metabolic syndrome; long-term effects secondary to cancer therapy in children; cardiovascular complications; cancer survivor; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood chronic myelogenous leukemia; juvenile myelomonocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Metabolic Syndrome; Leukemia, Myelomonocytic, Juvenile; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
RATIONALE: Gathering information about how often metabolic syndrome occurs in young survivors of childhood leukemia who have undergone stem cell transplant may help doctors learn more about the disease and the long-term effects of leukemia treatment. It may also help improve the quality of life for future cancer survivors.

PURPOSE: This clinical trial is studying metabolic syndrome in adolescent and young adult survivors of childhood leukemia who have undergone stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the prevalence of metabolic syndrome in adolescent and young adult survivors of childhood leukemia who have undergone hematopoietic stem cell transplantation (HSCT) and compare the extent to which prevalence is higher in HSCT survivors than in age- and gender-matched population norms derived from the Third National Health and Nutrition Examination Survey (NHANES III).
* To evaluate the relationship between insulin resistance and risk factors associated with metabolic syndrome (e.g., hypertension, obesity, hyperinsulinemia, and dyslipidemia) as measured by euglycemic insulin clamp, fasting serum insulin, glucose, lipids (total cholesterol, triglycerides, LDL-C, and HDL-C), blood pressure and anthropometric measurements, and DEXA scan in these patients and compare to age- and gender-matched population norms.
* To assess the extent to which prevalent obesity and insulin resistance are correlated with other factors that have been identified in the causal pathway associated with the development of metabolic syndrome and that may be altered after HSCT, including growth hormone secretion, adipokines (adiponectin and leptin), and inflammatory mediators (interleukin-6, tumor necrosis factor-α, and C-reactive protein).
* To evaluate the association of metabolic syndrome and early signs of impaired endothelial function and cardiovascular changes.
* To evaluate health behaviors related to prevention of cardiovascular disease, diabetes, and obesity, including a physical activity assessment, a dietary assessment, and a health knowledge assessment that will be used in the analyses of metabolic syndrome, growth hormone deficiency, and indicators of cardiovascular disease.

OUTLINE: Patients are stratified according to post-transplant follow-up period (2-9 years vs 10-15 years vs > 15 years).

Patients and their siblings undergo physical examination, a review of medical and family history, and blood pressure and anthropometric measurements. Patients and their siblings also undergo blood sample collection for laboratory studies (including analysis of C-reactive protein and CBC; lipid profile and triglycerides; leptin and adipokines; free thyroxine, TSH, IGF1, IGF3, and LH; and estradiol [females] or testosterone [males]); urine sample collection for microalbumin determination; and other study procedures (including euglycemic insulin clamp study; body composition and bone density [DEXA] study; bone-age x-ray [for patients < 18 years of age]; and vascular studies). Patients also undergo growth hormone stimulation testing.

Patients and their siblings complete questionnaires about their physical activity, dietary habits, and health knowledge.

PROJECTED ACCRUAL: A total of 193 childhood leukemia survivors and 193 healthy siblings will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Survivor of childhood leukemia, meeting all of the following criteria:

    * 21 years of age and under at diagnosis
    * Has undergone hematopoietic stem cell transplantation (HSCT) at Fairview University Medical Center or Fred Hutchinson Cancer Research Center ≥ 2 years ago
    * Disease in remission
  * Healthy sibling of a childhood leukemia survivor

PATIENT CHARACTERISTICS:

* Not pregnant
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 9 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Childhood leukemia survivors and healthy siblings, 9-21 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2005-04; Primary Completion 2011-07 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Comparison of the prevalence of metabolic syndrome in adolescent and young adult survivors of childhood leukemia who have undergone hematopoietic stem cell transplantation (HSCT) with age- and gender-matched controls | ≥2 years post-HSCT
Comparison of insulin resistance in patients with age- and gender-matched controls | ≥2 years post-HSCT
Correlation between insulin sensitivity and risk factors associated with metabolic syndrome | ≥2 years post-HSCT
Influence of time since transplant on insulin resistance | ≥2 years post-HSCT
Peak growth hormone secretion in patients with insulin resistance and in those without | ≥2 years post-HSCT
Growth hormone deficiency in patients with metabolic syndrome and in those without | ≥2 years post-HSCT
Association of interleukin-6, tumor necrosis factor-α, C-reactive protein, and leptin with insulin resistance and central obesity | ≥2 years post-HSCT
Correlation of adiponectin with insulin resistance and central obesity | ≥2 years post-HSCT
Differences in markers for endothelium dysfunction and early indicators of cardiovascular disease | ≥2 years post-HSCT
Difference in important health behaviors related to obesity and cardiovascular disease between patients with metabolic syndrome and those without | ≥2 years post-HSCT

CONTACTS AND LOCATIONS:
Overall Officials: K S Baker, MD, MS, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Clinical Research Center - Seattle Children's Hospital, Seattle, Washington, United States